CLINICAL TRIAL: NCT05472896
Title: TACE With Dicycloplatin（TP21） in Patients With Unresectable Hepatocellular Carcinoma: an Open, Parallel-controlled,Multicenter Randomized Phase III Trial
Brief Title: TACE With Dicycloplatin(TP21) in Unresectable HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gao-jun Teng (Other)
Responsible Party: Sponsor-Investigator, Gao-jun Teng, Clinical Professor, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TP21-TACE
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — diammine(1,1-cyclobutanedicarboxylate)platinum(II); Epirubicin

STUDY DESIGN:
Intervention Model Description: an open, parallel-controlled, multicenter randomized trial
Who Masked: Outcomes Assessor
Masking Description: the independent review committee (IRC) was used to evaluate the efficacy, and the readers reviewed the imaging data in a blinded state to make efficacy judgments. The following information was blinded to independent readers: subject's name, date of birth, personal information such as subject's initials, date of examination, statistical grouping, name of study unit, lesion selected by study unit for tumor evaluation, study Unit-determined tumor response and imaging reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTACE with TP21 (Experimental): In experimental groups, the dosage of dicycloplatin (TP21) was based on the body surface area (550 mg/m2) according to previous research. If grade III or above myelosuppression was observed, an adjusted dose of 450 mg/m2 was then considered, or the patient was removed from the group at the investigator's discretion.The volume ratio of lipiodol to dicycloplatin aqueous solution was 1:1.The volume of lipiodol used was calculated by the size and vascularity of the tumor, within 20 mL. Standardized gelatin sponge particles of 150-350 μm or 350-560 μm in diameter were injected following embolization with ethiodized oil-chemoembolic emulsion.
  Interventions: Procedure: cTACE; Drug: Dicycloplatin (TP21)
- cTACE with epirubicin (Active Comparator): the dosage of epirubicin was determined according to the tumor size, and the maximum dose was limited to 40 mg. The volume ratio of lipiodol to epirubicin aqueous solution was 2:1. The volume of lipiodol used was calculated by the size and vascularity of the tumor, within 20 mL. Standardized gelatin sponge particles of 150-350 μm or 350-560 μm in diameter were injected following embolization with ethiodized oil-chemoembolic emulsion.
  Interventions: Procedure: cTACE; Drug: Epirubicin

INTERVENTIONS:
Procedure: cTACE — transcatheter arterial chemoembolization with
Drug: Dicycloplatin (TP21) — the dosage of dicycloplatin was based on the body surface area (550 mg/m2) according to previous research. The volume ratio of lipiodol to dicycloplatin aqueous solution was 1:1. The volume of lipiodol used was calculated by the size and vascularity of the tumor, within 20 mL.
  Arms: cTACE with TP21
Drug: Epirubicin — the dosage of epirubicin was determined according to the tumor size, and the maximum dose was limited to 40 mg. The volume ratio of lipiodol to epirubicin aqueous solution was 2:1. The volume of lipiodol used was calculated by the size and vascularity of the tumor, within 20 mL.
  Arms: cTACE with epirubicin

SUMMARY:
To evaluate the effectiveness and safety of TP21 injection for TACE in treatment of hepatocellular carcinoma:

1. Primary efficacy endpoint: progression-free survival (PFS), which will be assessed by the Independent Review Committee according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST).
2. Secondary efficacy endpoints: PFS, objective response rate (ORR), disease control rate (DCR), overall survival (OS), time to progression (TTP), 1-year progression-free survival, 1-year survival and 2-year survival assessed by the investigator.

DETAILED DESCRIPTION:
TP21 injection is a supramolecular compound that has completed early pharmacological and toxicological preclinical studies, as well as phase I and II clinical studies. Data from previous studies showed that TP21 injection has significant advantages over traditional platinum-based drugs in terms of broad spectrum, low toxicity, high efficacy and low drug resistance etc. The results of the Phase II TACE clinical exploratory study in hepatocellular carcinoma showed a trend for TP21 alone to be significantly better than epirubicin alone, and due to the small sample size, the available data were insufficient to demonstrate obvious advantage of this drug. Now, a confirmatory phase III clinical study of TACE for hepatocellular carcinoma is needed, which may continue to adopt the main design of the phase II clinical trial, in a single agent comparison form: all the subjects will be randomized 1:1 into TP21+lipiodol group (trial group), and epirubicin hydrochloride+lipiodol group (control group) to receive TACE treatment of either "TP21+lipiodol" or "epirubicin hydrochloride+lipiodol". TACE treatment should be carried out for no more than 3 times in half a year to no more than 5 times within 1 year, and about 332 subjects will be enrolled, 166 for the trial group and the control group each.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older, and life expectancy ≥ 3 months;
2. histopathologically or clinically confirmed HCC;
3. Child-Pugh class A or B liver function (≤7 level), Eastern Cooperative Oncology Group performance status (PS) score of 0, 1 or 2；
4. China Liver Cancer stage IIb, IIIa (only Cheng's classification type I:portal vein tumor thrombus invading the portal vein branches of the liver lobe or liver segment) , and Ib, 2a patients who can be surgically removed, but are unable or unwilling to undergo surgery due to other reasons (such as advanced age, severe liver cirrhosis, etc.);
5. at least one lesion measurable by modified Response Evaluation Criteria in Solid Tumors for HCC (mRECIST);
6. no history of TACE or tumor recurrence after curative-intent therapy (i.e., surgical resection or ablation);
7. No blood transfusion and blood products, no use of granulocyte colony-stimulating factor (GCSF) and other hematopoietic stimulating factors within 2 weeks before screening; Hemoglobin ≥ 80g/L；Platelet count ≥ 60×10^9 /L; White blood cell count ≥ 3×10^9/L; Alanine aminotransferase ≤ 3 times the upper limit of normal; Aspartate aminotransferase ≤ 3×times the upper limit of normal; Serum creatinine Cr ≤ 1.5×times the upper limit of normal;

Exclusion Criteria:

1. allergic to platinum or iodine products or epirubicin and related excipients;
2. diffuse HCC (whole liver tumor burden ≥ 70%),and the hepatocellular carcinoma is hypovascular;
3. first-order branches and distant of the portal vein tumor thrombus;
4. Liver function classification is Child Pugh C;
5. Invasion of left and right hepatic duct, common hepatic duct, cystic duct and common bile duct;
6. The tumor has severe arteriovenous shunt, which the investigator judges may affect the efficacy of TACE; or there is extrahepatic metastasis;
7. Patients with other tumors, except for thyroid tumors and skin carcinoma in situ that have been cured, early cervical cancer;
8. Have a history of gastrointestinal bleeding or a marked tendency to gastrointestinal bleeding within 6 months before randomization;
9. Uncorrectable abnormal coagulation function or bleeding tendency;
10. received other antitumor therapies within the past 4 weeks (e.g., chemotherapy, radiotherapy, immunotherapy,Chinese medicine with antitumor effect), or received the above anti-tumor drugs within 5 half-lives;
11. received immunotherapy, targeted therapy or radiotherapy for intrahepatic tumors
12. have received an organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by Independent Review Committee | Up to ~1 years
  Progression-free survival (PFS) by Independent Review Committee (IRC) according to the Modified Response Evaluation Criteria in Solid Tumors (mRECIST).

SECONDARY OUTCOMES:
Progression-free survival (PFS) by investigator | Up to ~1 years
  Progression-free survival (PFS) by investigator according to the Modified Response Evaluation Criteria in Solid Tumors (mRECIST).
Objective Response Rate (ORR) | Up to ~1 years
Disease Control Rate (DCR) | Up to ~1 years
Overall Survival (OS) | Up to ~3 years
Time To Progress (TTP) | Up to ~3 years
1 year progression-free survival rate | Up to ~1 years
1 year survival rate | Up to ~1 years
2 year survival rate | Up to ~2years

OTHER OUTCOMES:
Adverse event/ serious adverse event | Up to ~2years

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, Doctor, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No